CLINICAL TRIAL: NCT03104933
Title: Proadrenomedullin and Copeptin as Predictors of Vasopressor Requirements and Volume Resuscitation in Patients With Septic Shock
Brief Title: Proadrenomedullin and Copeptin in Patients With Septic Shock
Acronym: proADM
Status: Completed | Type: Observational
Sponsor: Spanish Network for Research in Infectious Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 0530-N-16
Record Dates: First submitted 2017-03-20; First posted 2017-04-07 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2019-06

CONDITIONS: Septic Shock
Keywords: Proadrenomedullin; Copeptin; Vasopressors; Septic Shock
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with septic shock: patients in septic shock admitted to the ICU

SUMMARY:
This study evaluates the usefulness of pro-adrenomedullin (precursor of a vasodilatory peptide involved in septic shock pathogenesis) and copeptin (a stable peptide of the arginine vasopressin precursor) to predict, at the moment of septic shock diagnosis or their changes at 6 hours, the vasopressor requirements (measured by inotropic index and vasopressor dependency ratio) and volume requirement for resuscitation.

DETAILED DESCRIPTION:
Physiologically, adrenomedullin has a potent and prolonged vasodilatory effect. In both experimental animals and humans, the intravenous administration of ADM induces a marked and prolonged hypotension. Serum ADM levels are elevated in patients with septic shock. In fact, ADM seems to be one of the main mediators involved in hypotension that these patients present.

ADM is not stable in plasma due to its short half-life and rapid binding to receptors. ADM levels can be measured indirectly by determining proadrenomedullin (proADM) which is a more stable molecule and whose levels are reflected in the plasma of ADM.

Copeptin is released primarily in response to changes in serum osmolarity or blood volume by increasing peripheral vascular resistance and blood pressure.

Copeptin is elevated in patients with shock of different etiologies such as hemorrhagic shock or septic shock.

It is not defined in what situations and at what moment an invasive monitoring of the cardiac output and the different hemodynamic variables that reflect the preload and afterload in patients with septic shock should be performed. In fact, there is great variability in the management and treatment of patients with sepsis and septic shock, which includes the selection of patients who require invasive monitoring and the time of onset.

Having a biomarker or the combination of biomarkers that allow early determination of which patients will evolve poorly with the development of a shock that requires volume in large quantities and high doses of vasopressors will allow identifying a subgroup of patients that should be performed early hemodynamic monitoring and intensify medical treatment to try to reverse these severe hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Diagnosis of septic shock
* Obtaining written informed consent.

Exclusion Criteria:

* Initial dose of norepinephrine at ICU admission ≥ 0.6 mg / kg / min.
* Acute myocardial infarction in the previous month.
* History of pituitary surgery.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-07-01; Primary Completion 2019-09-30 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Levels of proADM as predictor of vasopressor requirements | the first 72 hours.
  measured by index inotropic and vasopressor dependency ratio) and fluid requirement
Levels o Copeptin as predictor of vasopressor requirements (measured by index inotropic and vasopressor dependency ratio) and fluid requirement | the first 72 hours.
  measured by index inotropic and vasopressor dependency ratio) and fluid requirement

SECONDARY OUTCOMES:
Levels of proADM and Copeptin as predictors of organ dysfunction | 28 days
  SOFA scale
Levels of proADM and Copeptin as predictor of 28-day mortality rate | 28 days
  Mortality
Levels of proADM and Copeptin as predictors of lactate clearance | 6 hours
  Lactate clearance

CONTACTS AND LOCATIONS:
Overall Officials: José Garnacho-Montero, MD, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- José Garnacho-Montero, Seville, Spain

IPD SHARING:
Plan to Share IPD: No